CLINICAL TRIAL: NCT01339533
Title: Airway Pressure Release Ventilation (APRV) vs. Conventional Volume Control Mechanical Ventilation for Patients With Respiratory Failure Requiring Invasive Mechanical Ventilator Support
Brief Title: Airway Pressure Release Ventilation (APRV) Versus AC/VC Conventional Ventilation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Eliotte L. Hirshberg, Principal Investigator, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APRV1015758
Record Dates: First submitted 2010-04-19; First posted 2011-04-20 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Failure; Acute Lung Injury (ALI); Acute Respiratory Distress Syndrome (ARDS)
Keywords: ALI; ARDS
MeSH Terms: conditions — Respiratory Insufficiency; Acute Lung Injury; Respiratory Distress Syndrome | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- APRV ls (Experimental): APRV low stretch will titrate Plow to maintain release volumes between 4 and 8 cc/kg.
  Interventions: Device: Mechanical Ventilation
- AC/VC Conventional Ventilation (Active Comparator): Standard volume control ventilation with the ARDS Net protocol.
  Interventions: Device: Mechanical Ventilation
- APRV h (Experimental): APRV Habashi protocol which sets Plow equal to 0.
  Interventions: Device: Mechanical Ventilation

INTERVENTIONS:
Device: Mechanical Ventilation — Patients who experience problems breathing and require assistance in breathing are placed on a machine that delivers air to the lungs through a tube through the vocal cords. This study is testing 3 protocols for that machine.

SUMMARY:
APRV mode of ventilation will result in an improved partial pressure of arterial oxygenation/ fraction of inspired oxygen (P/F ratio) on day 3 of mechanical ventilation. Sub hypotheses: APRV will be associated with a reduced amount of sedation used during the ICU stay in patients with respiratory failure. APRV will be associated with a reduction in the amount of vasoactive medication used for blood pressure support in patients with respiratory failure.

DETAILED DESCRIPTION:
This prospective un-blinded randomized trial will follow patients with respiratory failure and ALI/ARDS who require invasive mechanical ventilation in select ICUs. Patients will be allocated to respiratory support with either APRV mode or volume control (AC) mode of mechanical ventilation. Qualifying patients will be randomized by permuted block randomization within 24 hours of admission to the ICU. Identical ventilation and oxygenation thresholds will be utilized to guide titration of each ventilator protocol. Patients will remain on the assigned mode of ventilation until they are extubated and discharged from the ICU.

Procedures for treatment evaluation include daily monitoring of the Ventilator protocol in each arm. Clinical coordinator and study respiratory therapist will perform 2 daily checks of the study patients to determine compliance with the protocol and if patient meets weaning criteria. The previously published ARDS Network continuous positive airway pressure (CPAP) weaning protocol will be used for all patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic respiratory failure requiring mechanical ventilation for >24 hours.

Exclusion Criteria:

* Age under 18
* Severe chronic obstructive lung disease
* Patients in whom the only indication for mechanical ventilation is airway protection from poor neurological status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
P/F Ratio on Day 3 of Mechanical Ventilation | Day 3
  Our first objective is to measure and compare the partial pressure of oxygen in the artery to the inspired oxygen ratio (P/F ratio) on day 3 of mechanical ventilation. We will also collect and compare common variables used to evaluate lung injury and severity of respiratory failure in both groups. These variables and markers include: the Oxygenation index (OI) and standard blood gas parameters (PH, PaCO2 and PaO2).

SECONDARY OUTCOMES:
Amount/Duration of Sedative & Vasoactive Medication | Up to ICU discharge
  Our second objective is to compare the amount and duration of sedative medication and vasoactive medication per patient per/day required in each group. Duration of vasoactive medications and sedation (# of days) and quantitative amounts per kilogram will be compared. Measurements will include Mean Arterial Blood Pressure (MAP), Central venous pressure (CVP), and daily fluid balance between patients on AC and APRV.
Evaluate Feasibility & Clinical Compliance with 2 APRV Paper Protocols. | Up to ICU discharge
  Our third objective is to evaluate the feasibility of 2 previously developed APRV paper protocols (APRVa and APRVb) and document the clinician compliance with each paper APRV protocol. We will also track common events associated with mechanical ventilation. The incidence of pneumothorax defined as any ventilator-barotrauma resulting in chest tube placement, will be carefully followed.

CONTACTS AND LOCATIONS:
Overall Officials: Eliotte Hirshberg, MD, Principal Investigator — IHC Health Services, Inc., Dba: Intermountain Medical Center
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - LDS Hospital, Salt Lake City, Utah